CLINICAL TRIAL: NCT06264999
Title: Gait Analysis, Stair Performance and CT-based Micromotion Analysis in Robotic Assisted Total Knee Arthroplasty Comparing Bi-cruciate Retaining vs Cruciate Retaining Implants: A Single Centre Patient-blinded Randomized Controlled Trial
Brief Title: Robotic Assisted Knee Arthroplasty - Retain the Anterior Cruciate Ligament or Not
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to implant-related factors, forced to terminate the planned study
Sponsor: St. Olavs Hospital (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 427976
Record Dates: First submitted 2023-12-28; First posted 2024-02-20 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Arthritis Knee; Arthroplasty; Gait Analysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Journey II CR (Active Comparator): Implantation of Journey II CR sacrificing the anterior cruciate ligament.
  Interventions: Device: Journey II CR
- Journey II XR (Active Comparator): Implantation of Journey II XR retaining the anterior cruciate ligament.
  Interventions: Device: Journey II XR

INTERVENTIONS:
Device: Journey II CR — Implantation of Journey II CR Crucite Retaining Knee
  Arms: Journey II CR
Device: Journey II XR — Implantation of Journey II XR Bi Cruciate Retaining Knee
  Arms: Journey II XR

SUMMARY:
The goal of this clinical trial is to compare the function of the knee after retaining or sacrificing the anterior cruciate ligament in robotic assisted knee arthroplasty.

The main questions it aims to answer are:

Does retaining the anterior cruciate ligament improve postoperative gait? Participants will perform

* Gait analysis
* Stair performance test
* CT based Micromotion analysis of the implant micromovement

DETAILED DESCRIPTION:
A randomized controlled clinical trial intended to compare walking function and movement of the prosthesis after robot-assisted knee replacement surgery with two knee replacement designs; One prosthesis is preserving the anterior cruciate ligament (Smith+Nephew Journey II XR) and the other is sacrificing the anterior cruciate ligament (Smith+Nephew Jourrney II CR).

It is common to remove anterior cruciate ligament during knee replacement surgery. There is speculation about this weakens the balance in the operated knee and whether this can explain some of the problems that up to 20% experience after knee replacement surgery.

Preservation of the anterior cruciate ligament during knee replacement surgery may provide a more natural movement and better balance in the operated knee, and this in turn could provide increased patient satisfaction.

Previous studies have shown that knee replacement surgery where the anterior cruciate ligament is preserved has an increased incidence of per- and postoperative complications and reduced implant survival. Robot assisted navigation in knee arthroplasty surgery has shown the possibility of increased precision and accuracy when implanting the knee prostheses, and therefore might provide increased satisfaction when performing elective knee prosthetic surgery with robotic assistance and at the same time preserving the anterior cruciate ligament without an increased risk of complications.

In this study, postoperative function is assessed by looking at whether the walking pattern has normalized.

Gait analyses with comparison of the two groups is carried out both before surgery and 2, 6 and 12 months after surgery.

Primary endpoint is self-selected walking speed at 12 months follow-up. Secondary endpoints include other gait analysis parameters, result of stair test, as well as patient-reported pain, satisfaction and function (NRS, EQ-5D-5L, KOOS-PS, IKSS, FJS-12), knee mobility, stability, and hip-knee-ankle angle.

Complications related to the surgery or the course afterwards is noted. The study will also compare the movement of the prosthetic components in relation to the skeleton over a period of 2 years using a CT based micro motion analysis method (CT-RSA) making it possible to assess implant migration over time.

Increased movement can predict early loosening of the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Severe osteoarthritis Ahlbäck grade 3 or 4 affecting 2-3 compartments
* Ability to preoperatively walk 30 m independently without support before surgery
* Ability to give written consent.
* CPAK (Coronal Plane alignment of the Knee) I, II or III

Exclusion Criteria:

* Previous cruciate ligament surgery in affected knee
* Previous osteotomy in affected knee,
* Posttraumatic arthritis in affected knee
* History of infectious arthritis
* Rheumatoid arthritis
* Significant preoperative varus or valgus deformity >15º
* Evidence of damaged Anterior Cruciate Ligament and/or Posterior Cruciate Ligament
* Flexion contracture > 10 º, - Planning reveals the need for a complex implant ( stem, augment or higher level of constraint).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Preferred walking speed (meter/minute) after surgery | twelve months after surgery.
  Evaluation of gait with preferred walking speed (meter/minute) measured on a electronic walkway system
CT-RSA measured maximum total point of motion(MTPM) | 6,12 and 24 months after surgery
  CT-RSA measured maximum total point og motion(MTPM)in millimeters and rotation of the implant in degrees compared to baseline value

SECONDARY OUTCOMES:
evaluation of max walking speed(m/minute) | twelve months after surgery.
  Assesment of maximum walking speed(meter/minute) measured on a electronic walkway system
stride length(cm) | twelve months after surgery.
  Assesment of stride length (centimeters) measured on a electronic walkway system
step length in mid stance phase (cm) | twelve months after surgery.
  Assesment of step length(centimeters) in mid stance phase measured on a electronic walkway system
single leg support time(s) | twelve months after surgery.
  Assesment of single leg support time(seconds) measured on a electronic walkway system
double-leg support time(s) | twelve months after surgery.
  Assesment of double leg support time (seconds) measured on a electronic walkway system
stair performance(s) | twelve months after surgery.
  A 11-step stair ascend/descend test (STTotal-11) measures the time(seconds) it takes a subject to ascend and descend a flight of 11 steps (each step 17 cm high and 30 cm deep).
Rating pain using NRS (Numeric Rating Scale). | twelve months after surgery.
  NRS is a pain screening tool used to assess pain severity at that moment in time using a 0-10 scale, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable
KOOS-PS (Knee Injury and Osteoarthritis Outcome score) | twelve months after surgery.
  The KOOS-PS is a derivative of the Knee Injury and Osteoarthritis Score (KOOS). The KOOS-PS tool is intended to attain a feasible, short measure of physical function with interval level properties to assess the patient's opinion about their knee and associated problems.
  It measures Function (rising from sitting, bending to floor, putting on socks/stockings, rising from bed) and Sports (squatting, kneeling, twisting/pivoting) subscales. Items are scored from 0 to 4 and summed to give a raw score from 0 to 28, with lower scores representing higher levels of functional status.
Clinical evaluation of range of motion . | twelve months after surgery.
  Measure how much the knee will bend and extend in degrees both passive and active.
  Measure the Anterio-Posterior and Medio-Lateral stability i millimeters
Rating outcome using EQ-5D-5L(European quality of life index version 5D-5L), | twelve months after surgery.
  EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on scale that describes the degree of problems in that area (i.e. I have no problems walking about, slight problems, moderate problems, severe problems, or unable to walk). This tool also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.
IKSS (International Knee Society System knee and function score) | twelve months after surgery.
  Knee Society Clinical Rating System (KSS) provides a objective scoring system to rate the knee and patient's functional abilities before and after total knee arthroplasty.
  It has a Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee condition
FJS-12 (Forgotten Joint score) | twelve months after surgery.
  Forgotten Joint Score (FJS) is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment.
  The Forgotten Joint Score consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities
Clinical evaluation of Anteroposterior stability. | twelve months after surgery.
  The anterior-posterior (AP) stability of the knee is an important aspect of functional performance and is measured in millimeters
Clinical evaluation of Mediolateral stability. | twelve months after surgery.
  Mediolateral stability is measured in degrees and evaluated in 3 groups (Group 1: <5°, Group 2: 6°-9°, Group 3: ≥10°

OTHER OUTCOMES:
A long leg X-Ray identifying outliers with Hip Knee Ankle angle Varus <-3 ºor Valgus >3 º | 8 weeks
  Examination of long leg radiographs measuring the Hip-Knee Ankle angle in degrees
Presence of eminence fractures | 2 days postoperatively
  Examination of postoperative radiographs evaluating the presence of eminence fractures

CONTACTS AND LOCATIONS:
Overall Officials: Tina Strømdal-Wik, MD, PhD, Study Director — <St Olav- NTNU?
Locations (1):
- St.Olavs Hospital, Trondheim, Trøndelag, Norway